CLINICAL TRIAL: NCT00523640
Title: A Phase II Trial of Gemcitabine, Capecitabine, and Bevacizumab in Metastatic Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Too slow accrual
Sponsor: University of Chicago (Other)
Collaborators: Genentech, Inc. (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13662A
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Results first posted 2011-12-22 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-01

CONDITIONS: Carcinoma, Renal Cell
Keywords: metastatic; renal cell; kidney; neoplasm
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis; Neoplasms | interventions — Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- I (Experimental): Combination of gemcitabine, capecitabine, and bevacizumab
  gemcitabine 1000 mg/m^2 d1, 8, capecitabine 1000 mg (flat dose) po bid d1-14, and bevacizumab 15 mg/kg d 1, on a 21 day cycle
  Interventions: Drug: combination of gemcitabine, capecitabine, and bevacizumab

INTERVENTIONS:
Drug: combination of gemcitabine, capecitabine, and bevacizumab — gemcitabine 1000 mg/m^2 d1, 8, capecitabine 1000 mg (flat dose) po bid d1-14, and bevacizumab 15 mg/kg d 1, on a 21 day cycle

SUMMARY:
The purpose of this study is to find out what effects (good and bad) the combination of the chemotherapy drugs gemcitabine, capecitabine, and bevacizumab has on a patient and kidney cancer.

DETAILED DESCRIPTION:
* to determine the objective response rate and estimate the time to progression of combination gemcitabine, capecitabine, and bevacizumab in patients with metastatic clear cell renal cell cancer;
* to determine survival of combination gemcitabine, capecitabine, and bevacizumab in patients with metastatic cell renal cell cancer;
* to determine the toxicity of combination gemcitabine, capecitabine, and bevacizumab in patients with metastatic renal cell cancer;
* to collect baseline serum and plasma samples for exploration of possible prognostic and predictive markers

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic clear cell renal cell cancer
* Measurable disease
* Age 18 or older
* ECOG performance status of 0 - 1
* Blood pressure less than 140/90 on 2 separate occasions not more than 6 weeks prior to enrollment and not less than 24 hours apart
* Normal organ function
* Women of child-bearing potential and men must agree to use adequate contraception
* Ability to understand and the willingness to sign a written informed consent document and to follow all required study procedures

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not have had prior treatment with pyrimidine analogs or VEGF binding agents
* Patients may not be receiving any other investigational or therapeutic agents
* Patients may not be receiving therapeutic anticoagulation with warfarin, its congeners, heparin, low molecular weight heparinoids, specific thrombin inhibitors, or other similar agents Patients receiving low dose coumadin (1 mg daily) for central line patency are eligible
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to treatment start, or anticipation of need for major surgical procedure during the course of the study Fine needle aspirations or core biopsies within 7 days prior to treatment start are acceptable
* Serious, nonhealing wound, ulcer, or bone fracture
* Evidence of bleeding diathesis or coagulopathy
* Patients with known brain metastases
* Uncontrolled intercurrent illness
* Pregnant women
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Stadler, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 patients were enrolled in the trial between March 2005 and May 2008
Groups:
- Combination of Gemcitabine, Capecitabine, and Bevacizumab: combination of gemcitabine, capecitabine, and bevacizumab
Period: Overall Study
Arm/Group | Combination of Gemcitabine, Capecitabine, and Bevacizumab
Started | 30
Completed | 29 (1 patient died before starting treatment)
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Combination of Gemcitabine, Capecitabine, and Bevacizumab
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 58 [36 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29
Performance Status [Number; unit: participants] — ECOG performance status Scores on a scale Range 0-5, higher is worse
  participants
    0 | 5
    1 | 23
    2 | 1
Number of metastatic disease sites [Number; unit: participants]
  1 | 2
  2 | 6
  3 or more | 21
Tumor histology [Number; unit: participant]
  Clear cell | 23
  Poorly differentiated/unclassified | 6
Fuhrman grade [Number; unit: participants] — An important factor used to assess renal cell carcinoma is its Fuhrman grade. This scale refers to how closely the cancer cells look like normal kidney cells under a microscope. The Fuhrman grading system ranks tumor cells on a scale of 1 through 4 and is a prognostic scale. 1 represents the best prognosis and 4 the worst. Grade 1 tumor cells look similar to normal kidney cells. Grade 1 cancers typically grow and spread slowly and most often have a good prognosis. Grade 4 tumor cells look quite different from normal kidney cells and have a worse prognosis.
  participants
    1 | 0
    2 | 2
    3-4 | 21
    Unknown | 6
Prognostic risk group [Number; unit: participants]
  Favorable | 7
  Intermediate | 19
  Poor | 3
Prior therapy-Nephrectomy [Number; unit: participants]
  Yes | 24
  No | 5
Prior therapy-Radiotherapy [Number; unit: participants]
  Yes | 15
  No | 14
Prior therapy-Cytokine therapy [Number; unit: participants]
  Yes | 8
  No | 21
Prior therapy-Oral Vascular Endothelial Growth Factor (VEGF) receptor kinase inhibitor [Number; unit: participants]
  Yes | 20
  No | 9

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Per RECIST Criteria (V1.0) using standard cross-sectional CT scanning: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Response (R)= CR + PR.
Time Frame: 12 weeks
Measure: Number; unit: proportion
Arm/Group | Combination of Gemcitabine, Capecitabine, and Bevacizumab
Number analyzed (Participants) | 29
proportion | 0.24 [0.10 to 0.44]
Statistical Analysis 1: Comparison: Combination of Gemcitabine, Capecitabine, and Bevacizumab; Test type: Superiority or Other; Proportion responding = 0.24, 95% CI 2-sided [0.10 to 0.44]

2. Primary Outcome: Progression-free Survival
Description: Progression is defined as a measurable increase in the sum of longest diameters of all target lesions, or unequivocable progression of non-target lesions, or the appearance of new lesions, since baseline
Time Frame: 60 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination of Gemcitabine, Capecitabine, and Bevacizumab
Number analyzed (Participants) | 29
months | 5.3 [3.9 to 9.9]

3. Secondary Outcome: Overall Survival
Description: Time from enrollment until death from any cause.
Time Frame: 60 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Combination of Gemcitabine, Capecitabine, and Bevacizumab
Number analyzed (Participants) | 29
months | 9.8 [6.2 to 14.9]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored over the course of treatment
Description: Reported are numbers of patients with grade 3 or higher toxicity National Cancer Institute Common Toxicity Criteria (version 3.0) were used to assess and report adverse events
Arm/Group | Combination of Gemcitabine, Capecitabine, and Bevacizumab
Serious Adverse Events (participants affected / at risk) | 5/29
Other Adverse Events (participants affected / at risk) | 20/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination of Gemcitabine, Capecitabine, and Bevacizumab (N=29)
Seizure (Nervous system disorders) | 1
Sepsis (Infections and infestations) | 1
Bowel perforation (Gastrointestinal disorders) | 1
Pulmonary Embolism/Deep Vein Thrombosis (Blood and lymphatic system disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Combination of Gemcitabine, Capecitabine, and Bevacizumab (N=29)
Leukopenia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 9
Anemia (Blood and lymphatic system disorders) | 4
thrombocytopenia (Blood and lymphatic system disorders) | 2
Hand foot syndrome (Skin and subcutaneous tissue disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Fatigue (General disorders) | 6
Nausea (Gastrointestinal disorders) | 2
Emesis (Gastrointestinal disorders) | 2

LIMITATIONS AND CAVEATS:
Trial was designed with a maximum target accrual of 55 patients. The trial was halted early because emerging data with VEGF inhibitors challenged clinical relevance of the study and availability of multiple therapies challenged accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes